CLINICAL TRIAL: NCT02494154
Title: Effects of Treatment With High Flow Nasal Cannulas on Respiratory Pattern and Work of Breathing Among Patients.
Acronym: HDWOBPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IUCPQ-HDWOBPT
Record Dates: First submitted 2015-06-04; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Conventional flow via nasal prongs (Active Comparator): Oxygen delivery via conventional nasal interface with flow adjusted to reach a target SpO2 according to the patient's condition.
  Interventions: Device: Oxygen delivery via conventional nasal mask
- High flow nasal cannulas 20L/min (Experimental): Oxygen delivery via high flow nasal cannulas (20L/min) with fraction of inspired oxygen (FiO2) adjusted to reach a target SpO2 according to the patient's condition.
  Interventions: Device: Airvo 2; Ficher and Paykel HealthCare
- High flow nasal cannulas 40L/min (Experimental): Oxygen delivery via high flow nasal cannulas (40L/min) with FiO2 adjusted to reach a target SpO2 according to the patient's condition.
  Interventions: Device: Airvo 2; Ficher and Paykel HealthCare
- High flow nasal cannulas 60L/min (Experimental): Oxygen delivery via high flow nasal cannulas (60L/min) with FiO2 adjusted to reach a target SpO2 according to the patient's condition.
  Interventions: Device: Airvo 2; Ficher and Paykel HealthCare

INTERVENTIONS:
Device: Airvo 2; Ficher and Paykel HealthCare — High flow nasal cannulas
  Arms: High flow nasal cannulas 20L/min; High flow nasal cannulas 40L/min; High flow nasal cannulas 60L/min
Device: Oxygen delivery via conventional nasal mask — Low flow of oxygen delivered through conventional nasal prongs
  Arms: Conventional flow via nasal prongs

SUMMARY:
This study evaluates the work of breathing among patients under various conditions of treatment with high flow nasal cannulas. Sixteen spontaneously breathing patients with respiratory failure (hypercapnic or hypoxemic) will be included. The design of this study is a cross over of four treatment periods with different flow settings.

DETAILED DESCRIPTION:
High flow oxygen therapy (HFOT) is a promising technique increasingly used in the management of acute respiratory failure. In hospitalised hypoxemic patients, recent clinical evidence showed that HFOT can reduce endotracheal intubation and reduce mortality. Physiologically, the HFOT causes a decrease in respiratory rate and minute-ventilation and may be associated with a decrease in PaCO2. It is possible that these effects are associated with decreased work of breathing, which could explain some of the benefits in terms of comfort and efficiency.

The objective of this research is to evaluate the impact of a wash-out of anatomical dead space by high flow nasal cannulas on respiratory parameters and on the work of breathing.

The investigators will evaluate the baseline status with conventional oxygen therapy methods (low flows), and then compare it with three different levels of high flow oxygen therapy in a randomised order. The primary endpoint will be the work of breathing.

ELIGIBILITY:
Inclusion Criteria:

Spontaneously breathing patients exhibiting a respiratory distress defined by a respiratory rate ≥ 20 breaths/min associated with

* either hypoxemia (SpO2<90% with O2≥3L/min) ;
* or hypercapnia (PaCO2>45 mmHg with a respiratory acidosis (pH<7,38).

Exclusion Criteria:

* Patients below 18yo, pregnant or breastfeeding women;
* Patients enrolled in another study excluding co-enrolment;
* History of ear nose and throat disease (i.e. surgery, epistaxis, trauma), eso-gastric disease (i.e. esophageal varices, digestive haemorrhage), rheumatologic or neurologic disease possibly interfering with the design of the study;
* Acute respiratory or cardiovascular disease contra-indicating the enrolment in the study protocol (i.e. acute coronary syndrome, pulmonary embolism, pneumothorax);
* Need for immediate intubation or for continuous noninvasive ventilation and/or recent (<6h) arterial blood gases showing a respiratory acidosis with a pH<7.30;
* Patient feeling nauseous or under recent fed condition (<1h).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Work of breathing | 15 minutes
  Work of breathing at the end of each period is calculated from the measurement of esophageal pressure and tidal volume (composite outcome)

SECONDARY OUTCOMES:
Esophageal pressure-time product | 15 minutes
  Measured at the end of each period
Tidal volume | 15 minutes
  Measured at the end of each period
Comfort of breathing | 15 minutes
  Subjective evaluation at the end of each period
Blood gases | 15 minutes
  Arterial or capillary blood gases at the end of each period
Dyspnea | 15 minutes
  Evaluation on a borg scale at the end of each period
Respiratory rate | 15 minutes
  Measured at the end of each period
Heart rate | 15 minutes
  Measured at the end of each period
End-tidal carbon dioxide | 15 minutes
  Measured at the end of each period
Oxygen saturation | 15 minutes
  Measured at the end of each period

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, MD, PhD, Study Director — Fondation IUCPQ
Locations (1):
- IUCPQ, Québec, Quebec, Canada